CLINICAL TRIAL: NCT06699602
Title: A Pilot Phase II Study of Neoadjuvant Cemiplimab + Fianlimab in Patients With Locally Advanced Clear Cell Renal Cell Carcinoma Undergoing Nephrectomy
Brief Title: A Study of Cemiplimab and Fianlimab in People With Clear Cell Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-329
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Renal Cell Carcinoma
Keywords: Cemiplimab; Fianlimab
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cemiplimab and Fianlimab (Experimental): All patients will be treated as follows: cemiplimab and fianlimab every 3 weeks for a total of 3 treatments, or until unacceptable toxic effects, overt disease progression, or withdrawal from study.
  Interventions: Drug: Cemiplimab; Drug: Fianlimab

INTERVENTIONS:
Drug: Cemiplimab — cemiplimab IV flat
Drug: Fianlimab — fianilmab IV flat

SUMMARY:
The researchers are doing this study to find out whether it is practical (feasible) to give cemiplimab and fianlimab before a nephrectomy and whether it causes any delays with surgery in people with kidney cancer. The researchers will also look at whether cemiplimab and fianlimab given before a nephrectomy is a safe and effective treatment approach and if there is a change in the size of the tumor following immunotherapy prior to planned surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of informed consent.
2. Patient must be able to provide informed consent, or a legal authorized representative (LAR) must be identified to provide consent in cases where the patient cannot.
3. Signed and dated IRB-approved Informed Consent Form
4. Patients must be planned for nephrectomy for high risk non-metastatic clear cell renal cell carcinoma.

   * Non-metastatic disease will be defined by no evidence of metastases other than regional lymphadenopathy as assessed by imaging of the chest, abdomen and pelvis with CT of the chest and MR of the abdomen/pelvis (CT abdomen/pelvis will suffice for those unable to undergo MR imaging).
   * 'High-risk non-metastatic' is defined as those patients with a 12-year probability of metastases of ≥ 40% as per an established pre-operative nomogram
5. Patients must undergo baseline biopsy to confirm clear cell histology prior to treatment initiation.
6. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Patients must have adequate organ and bone marrow function, defined by the following laboratory results obtained within 14 days prior to the first study treatment:

   i. ANC ≥ 1500 cells/μL (without granulocyte colony stimulating factor support within 2 weeks prior to Cycle 1, Day 1) ii. WBC counts ≥ 2500/μL and ≤ 15,000/μL without G-CSF iii. Absolute Lymphocyte count ≥ 500/μL iv. Platelet count ≥100,000/μL (without transfusion within 2 weeks prior to Cycle 1, Day 1) v. Hemoglobin ≥9.0 g/dL (without transfusion within 2 weeks prior to Cycle 1, Day 1) vi. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 3 X upper limit of normal (ULN). ALP ≤ 5 x ULN if patient has documented bone metastases.

vii. Serum bilirubin ≤ 1.5 x ULN. Patients with known Gilbert disease who have serum bilirubin level ≤ 2 x ULN may be enrolled.

viii. Creatinine ≤ 2.0 x ULN or Estimated Glomerular Filtration Rate (eGFR) ≥ 40mL/min using the CKD-EPI formula.

Exclusion Criteria:

1. Prior receipt of any systemic therapy for renal cell carcinoma.
2. Prior receipt of any immune checkpoint inhibitor therapy for any indication.
3. Inability to safely delay surgery by 9 weeks as per surgeon's discretion.
4. Patients who are receiving any other investigational agents.
5. History of allergic reactions or known hypersensitivity attributed to the active substances or to any of the excipients
6. History of severe hypersensitivity reaction to any monoclonal antibody.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring therapy, symptomatic congestive heart failure, unstable angina pectoris, or uncontrolled cardiac arrhythmia.
8. Patients with a history of myocarditis.
9. Patients with Troponin TnT or troponin I TnI > 2x institutional ULN at baseline.

   ° Patients with TnT or TnI levels between > 1 to 2x ULN are permitted if repeat levels within 24 hours are ≤ 1x ULN. If TnT or TnI levels are > 1 to 2x ULN within 24 hours, the subject may undergo a cardiac evaluation and be considered for treatment by the investigator based on the medical judgement in the patient's best interest.
10. Patients with active autoimmune disease or recent history (within 2 years) of autoimmune disease that might recur, which may affect vital organ function, or require immune suppressive treatment including systemic corticosteroids, should be excluded. These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as SLE, connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease. Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event).
11. Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of study drug administration. Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
12. Diagnosis of another malignancy within 2 years before first dose of study treatment, except for superficial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy.
13. Prior allogeneic stem cell transplant or solid organ transplant.
14. History or current evidence of significant (CTCAE grade ≥2) local or systemic infection (eg, cellulitis, pneumonia, septicemia) requiring systemic antibiotic treatment within 2 weeks prior to the first dose of trial medication.
15. Use of live vaccines against infectious disease (e.g. varicella) within 30 days of initiation of study therapy. Killed vaccinations (e.g. influenza) are allowed at any appropriate time before and during the study. If a patient intends to receive a COVID19 vaccine before the start of study drug, participation in the study should be delayed at least 1 week after any COVID-19 vaccination. During the treatment period, it is recommended to delay COVID-19 vaccination until patients are receiving and tolerating a steady dose of study drug. A vaccine dose should not be less than 48 hours before or after study drug dosing.
16. Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C virus (HBV or HCV) infection; or diagnosis of immunodeficiency that is related to, or results in chronic infection.

    * Patients with known HIV infection who have controlled infection (undetectable viral load on HIV RNA PCR) and CD4 count above 350 (either spontaneously or on a stable antiviral regimen) are permitted. For patients with controlled HIV infection, monitoring will be performed per local standards.
    * Patients with HBV (hepatitis B surface antigen positive; HBsAg+) who have controlled infection (serum HBV DNA PCR that is below the limit of detection and receiving anti-viral therapy for HBV) are permitted. Patients with controlled infections must undergo periodic monitoring of HBV DNA. Patients must remain on anti-viral therapy for at least 6 months after the last dose of cemiplimab.
    * Patients who are HCV antibody positive (HCV Ab+) who have controlled infection (undetectable HCV RNA by PCR, either spontaneously or in response to successful prior course of anti-HCV therapy) are permitted.
    * Patients with HIV or hepatitis must be reviewed by a qualified specialist (eg, infectious disease or hepatologist) managing this disease prior to commencing and regularly throughout the duration of their participation in the trial
17. Women with a positive serum beta-hCG pregnancy test at screening/baseline visit. If positive, pregnancy must be ruled out by ultrasound for patient to be eligible.
18. Breast-feeding women.
19. Women of childbearing potential (WOCBP) who are sexually active and are not willing to practice highly effective contraception prior to the first treatment, during the study, and for at least 6 months after the last dose. Highly effective contraceptive measures include:

    * stable use of combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal) or progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation initiated 2 or more menstrual cycles prior to screening;
    * intrauterine device; intrauterine hormone-releasing system;
    * bilateral tubal occlusion/ligation;
    * vasectomized partner (provided that the male vasectomized partner is the sole sexual partner of the WOCBP study participant and that the vasectomized partner has obtained medical assessment of surgical success for the procedure); and/or
    * sexual abstinence - Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drugs. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.
20. Male study participants with WOCBP partners are required to use condoms during the study and until 6 months after the last dose of study treatment unless they are vasectomized or practice sexual abstinence.
21. WOCBP must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the entire trial and until 6 months after last treatment.
22. All men must agree not to donate sperm during the trial and for 6 months after receiving the last therapy dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
response | 1 year
  will be evaluated in this study using the international criteria proposed by RECIST version 1.1. Changes in the largest diameter (unidimensional measurement) of the tumor lesion and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Martin Voss, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activites), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering West Harrison (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activites), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm